CLINICAL TRIAL: NCT00312286
Title: A Randomized, Placebo-Controlled Phase II Study of Multiple Dosing Regimens of Intravaginally Administered 851B Gel for the Treatment of Cervical High Risk HPV Infection
Brief Title: Efficacy of 851B Gel for Treating High-Risk Cervical Human Papillomavirus Infection in Women.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1547-851B; U1111-1127-5771 (Registry Identifier: WHO)
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Papillomavirus Infections
Keywords: Cervical Neoplasms; Drug Therapy; Human Papillomavirus; Cervical Human Papillomavirus; Cervical Dysplasia; Chemoprevention; High Risk Cervical Human Papillomavirus; Atypical Squamous Cells of Undetermined Significance; Low Grade Intraepithelial Lesions
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Atypical Squamous Cells of the Cervix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- 1 (Experimental)
  Interventions: Drug: 851B
- 2 (Experimental)
  Interventions: Drug: 851B
- 3 (Experimental)
  Interventions: Drug: 851B
- 4 (Experimental)
  Interventions: Drug: 851B
- 5 (Experimental)
  Interventions: Drug: 851B
- 6 (Experimental)
  Interventions: Drug: 851B
- 7 (Experimental)
  Interventions: Drug: 851B
- 8 (Placebo Comparator)
  Interventions: Drug: 851B
- 9 (Placebo Comparator)
  Interventions: Drug: 851B
- 10 (Placebo Comparator)
  Interventions: Drug: 851B
- 11 (Placebo Comparator)
  Interventions: Drug: 851B

INTERVENTIONS:
Drug: 851B — 851B 0.15% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 1
Drug: 851B — 851B 1.5% formulation, gel, topically, twice a week for 1 cycle.
  Arms: 2
Drug: 851B — 851B 1.5% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 3
Drug: 851B — 851B 3.0% formulation, gel, topically, once a week for 1 cycle.
  Arms: 4
Drug: 851B — 851B 3.0% formulation, gel, topically, once a week for 2 cycles.
  Arms: 5
Drug: 851B — 851B 3.0% formulation, gel, topically, twice a week for 1 cycle.
  Arms: 6
Drug: 851B — 851B 3.0% formulation, gel, topically, twice a week for 2 cycles.
  Arms: 7
Drug: 851B — 851B placebo-matching gel, topically, once a week for 1 cycle.
  Arms: 8
Drug: 851B — 851B placebo-matching gel, topically, twice a week for 1 cycle.
  Arms: 9
Drug: 851B — 851B placebo-matching gel, topically, once a week for 2 cycles.
  Arms: 10
Drug: 851B — 851B placebo-matching gel, topically, twice a week for 2 cycles.
  Arms: 11

SUMMARY:
The purpose of this study was to evaluate efficacy of 851B gel over a range of concentrations and dosing regimens on high-risk cervical human papillomavirus infection in women.

DETAILED DESCRIPTION:
Cervical cancer is caused by infection with specific genotypes of the human papillomavirus referred to as oncogenic or high-risk human papillomavirus. Current epidemiologic evidence suggests that 80% of sexually active women will become infected during their lifetime with human papillomavirus and 50% of these infections will be due to high-risk human papillomavirus. With US annual rates of cervical cancer now in the range of 13,000/year, a very substantial number of women are left with uncertainty regarding whether their infection will clear spontaneously or progress to cancer.

Subjects participating in this study were required to visit the clinic for approximately 15 or 16 visits, and maintain a diary of self-dosing and menstruation cycles. The total time of participation in this study was approximately 27 months.

ELIGIBILITY:
Inclusion Criteria:

* A female subject of childbearing potential who is sexually active using contraception.
* Subject is willing to abstain from all sexual contact involving her genitalia for at least 24 hours prior to and 24 hours after study drug administration.
* Subject must be neither pregnant nor lactating from Screening throughout the duration of the study.
* Subject has 1 of the following:

  * Menstruating with a stable cycle and has at least 21 non-bleeding days.
  * Amenorrheic (due to injectable or extended-cycle contraceptives).
* Subject is willing to refrain from using vaginal douche products during the treatment period and through the Follow-up Month 4 visit.
* Subject has a Pap test interpretation of either low-grade squamous intraepithelial lesions or atypical squamous cells of undetermined significance.
* Subject has a uterine cervical sample that is high-risk human papillomavirus positive.

Exclusion Criteria:

* The Subject has evidence of an uncontrolled, clinically significant medical condition as determined by the investigator.
* The Subject has a history of hemorrhagic diatheses or coagulopathy.
* The Subject has a history of toxic shock syndrome.
* The Subject has received any of the following medications in the timeframes listed below:

  * 851 (in any form) or an active (non-placebo) human papillomavirus vaccine at any time prior to the screening visit.
  * In the 4 weeks prior to the screening visit the subject has received:

    * Interferon therapy or other therapies that promote a proinflammatory immune state, including:

      * immunomodulators.
      * cytotoxic drugs.
      * drugs known to have major organ toxicity.
    * Used a vaginal douche 72 hours prior to the screening visit.
    * Received any investigational drug within 60 days of Study Day 1.
    * Used in the 2 weeks prior to Study Day 1:

      * oral or inhaled corticosteroids (>1000 mcg/day, fluticasone propionate >600 mg/day, or equivalent).
      * systemic steroids.
      * topical drugs to the anogenital area.
      * NuvaRing.
* The Subject has a history of hypersensitivity to any components of the gel formulation or to iodine.
* The Subject has given birth or has had a spontaneous or induced abortion within 2 months of Study Day 1.
* The Subject uses an intrauterine device, diaphragm, NuvaRing, or additional contraceptive foam or gel for birth control.
* The Subject has:

  * histology read as high-grade cervical intraepithelial neoplasia.
  * cytology read as high-grade squamous intraepithelial lesion.
  * cytology read as atypical glandular cytological abnormalities.
  * cytology read as atypical squamous cells - cannot exclude high grade.
  * cervical carcinoma of any type.
  * apparent endocervical involvement.
  * high-grade vulvar intraepithelial neoplasia.
  * high-grade vaginal intraepithelial neoplasia.
* If the limits of a cervical lesion cannot be readily visualized.
* If the limits of the transformation zone cannot be readily visualized.
* The subject has clinical evidence of a vaginal infection or sexually transmitted infection, other than cervical human papillomavirus infection at the Study Day 1 visit.
* The Subject has had a cervical biopsy within 1 month prior to the screening visit.
* The Subject has had any previous ablative or surgical treatment of the cervix within 3 months prior to the screening visit;
* The Subject has a history of alcoholism or substance abuse within 1 year or has current alcohol or substance abuse as assessed by the investigator.
* The Subject has tested positive for human immunodeficiency virus at the screening visit or has evidence of any other immunosuppressive disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 538 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Time to clearance of high-risk human papillomavirus infection. | At each visit

SECONDARY OUTCOMES:
Proportion of subjects with evidence of regression to normal cytology. | Screening Visit and Follow-up Visits (Months 6, 8, 14, 20, and 26).
Proportion of subjects with improvement in cervical lesions as rated by the investigator (measured by colposcopy). | At each visit
Proportion of subjects who develop histological evidence of cervical intraepithelial neoplasia. | Visits 1-3 as assigned by group
Time to progression of disease to precancer. | Visits 1-3 as assigned by group
Change in relative light units ratios relative to the positive control from Hybrid Capture 2® assay (semi-quantitatively assessing viral load). | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (93):
- United States (88):
  - Birmingham, Alabama
  - Enterprise, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Carmichael, California
  - Colton, California
  - San Diego, California
  - San Francisco, California
  - Santa Rosa, California
  - Colorado Springs, Colorado
  - Longmont, Colorado
  - Louisville, Colorado
  - Danbury, Connecticut
  - Groton, Connecticut
  - Aventura, Florida
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Evansville, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Marrero, Louisiana
  - Metairie, Louisiana
  - Detroit, Michigan
  - Paw Paw, Michigan
  - Chaska, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Reno, Nevada
  - Lebanon, New Hampshire
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Gallipolis, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Pottstown, Pennsylvania
  - West Reading, Pennsylvania
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Watertown, South Dakota
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Clarksville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sandy City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
  - Seattle, Washington
- Canada (4):
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Québec, Quebec
  - Toronto
- Rio Piedras, Puerto Rico